CLINICAL TRIAL: NCT07033416
Title: A Pilot Randomised Controlled Trial of Approach Bias Modification During Traetment for Cocaine Use Disorder
Brief Title: A Trial Of Approach Bias Modification Training During Treatment For Cocaine Use Disorder
Acronym: ABMCocaine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Collaborators: Monash University (Other)
Responsible Party: Principal Investigator, Doriana Losasso, Psych, Principal Investigator, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABMCocaine
Record Dates: First submitted 2025-06-05; First posted 2025-06-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-06

CONDITIONS: Training for Cocaine Use Disorder
Keywords: APPROACH BIAS MODIFICATION; RCT; COCAINE USE DISORDER
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABM+TAU (Experimental): Participants treated with the experimental training Approach Bias Modification (ABM), and the usual treatment (Treatment As Usual, TAU).
  Interventions: Behavioral: Approach Bias Modification; Behavioral: Treatment as usual
- TAU (Active Comparator): Participants treated with the usual treatment (Treatment As Usual, TAU).
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Approach Bias Modification — ABM is a computerised training aiming to train the participants to avoid drug-related images (by pushing a joystick which causes the image to disappear) and approach positive images (by pulling a joystick which causes the image to expand). Each training session lasts 15 minutes and it takes place once per week for 4 weeks.
  Arms: ABM+TAU
Behavioral: Treatment as usual — Participants receiving TAU are not trained to avoid drug-related images and approach positive images.

SUMMARY:
The goal of this clinical trial is to investigate if the intervention "Approach Bias Modification" (ABM) can low cocaine craving in people with Cocaine Use Disorder (CUD).

The main question this clinical trial aims to answer is how many days participants can be in abstinence from cocaine after 4 ABM sessions.

ABM is a computerised training aiming to train the participants to:

* avoid drug-related images by pushing a joystick which causes the image to disappear;
* approach positive images by pulling a joystick which causes the image to expand.

Researchers will compare participants treated with ABM to those who receive Treatment As Usual (TAU) condition to see if ABM training for CUD is more effective in increasing the number of abstinent days.

* Participants will attend 1 ABM session per week for a total of 4 sessions, each lasting 15 minutes.
* Both cocaine and non-cocaine positive images relative to the subjective values or interests (i.e. effects, sport, music, nature, work, etc.) are presented to the participant, in portrait or landscape orientation.
* Participants are instructed to push the joystick if the image is portrait-oriented (cocaine-related images) or to pull the joystick if it is landscape-oriented (positive images).
* At 1 and 3-month-follow up, participants will complete self-report questionnaires to measure abstinence days and describe the effect of ABM on cocaine use, dependence symptoms, and approach bias.

ELIGIBILITY:
Inclusion Criteria:

* participants must be aged at least 18 years;
* current DSM 5 TR Cocaine Use Disorder;
* sufficient Italian language proficiency to understand the participant information sheet, questionnaires and intervention task instructions;
* signed Consent form.

Exclusion Criteria:

Participants are excluded from participating if they have:

* neurological disorder or injury or brain trauma involving loss of consciousness for longer than 30 minutes;
* severe psychiatric disorder, as evaluated by clinical judgement;
* antipsychotic medication;
* intellectual disability;
* missing Informed Consent;
* planned absence from attendance through the training period (one month).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Abstinence days from cocaine after 4 Approach Bias Modification (ABM) training sessions | Urine analysis from enrollment to the end of treatment twice a week,in the first three weeks. TLFB at 1 and 3 months after the end of training.
  Abstinence days from cocaine measured by urine analysis and a self-report questionnaire (Timeline Follow-Back, TLFB) measuring frequency and quantity of cocaine use and route of administration.

SECONDARY OUTCOMES:
Operationalisation of continuous abstinence in participants trained with ABM, relative to TAU. | at 1 and 3 months after the end of training.
  Operationalisation of continuous abstinence is assessed by urine analysis and self-report questionnaires:
  • Craving Experience Questionnaire (CEQ): two 10-item scales, one measuring the frequency of cravings over a defined time period, and the other assessing the strength of the strongest cravings during this period.
Operationalisation of continuous abstinence in participants trained with ABM, relative to TAU | at 1 and 3 months after the end of training
  Severity of Dependence Scale (SDS): a continuous measure of psychological dependence on cocaine. A score of zero is assigned to no cocaine use during the past month.
Operationalisation of continuous abstinence in participants trained with ABM, relative to TAU. | at 1 and 3 months after the end of training
  Operationalisation of continuous abstinence is assessed by urine analysis and self-report questionnaires:
  Timeline Follow-back (TLFB): a measure of frequency and quantity of cocaine use and route of administration
Operationalisation of continuous abstinence in participants trained with ABM, relative to TAU. | at 1 month after the end of training
  Operationalisation of continuous abstinence is assessed by urine analysis and self-report questionnaires:
  Modified Stroop Task for Addiction (MST): a 0-to-100 scale measuring attention regulation and suppression of interference due to semantic incongruence or salience of addiction-related stimuli.
Operationalisation of continuous abstinence in participants trained with ABM, relative to TAU. | at 1 month after the end of training
  Operationalisation of continuous abstinence is assessed by urine analysis and self-report questionnaires:
  Modified Go/No-go Task for Addiction (MGNT): a measure of suppression of pre-potent responses and control of attention bias for salient stimuli associated with addiction-related.

CONTACTS AND LOCATIONS:
Overall Officials: Doriana Losasso, Principal Investigator — ASST Fatebenefratelli Sacco
Locations (1):
- Struttura Semplice Servizio Dipendenze, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No
At present ethics has not approved the sharing of IPD with researchers outside of the investigator team